CLINICAL TRIAL: NCT01024491
Title: A Parallel Randomized Double Blind Placebo Controlled Clinical Trial to Study the Efficacy and Safety of Paroxetine Daily Doses of 15 mg and 20 mg in the Treatment of Premature Ejaculation
Brief Title: Efficacy and Safety of Paroxetine Daily Doses of 15 mg and 20 mg in the Treatment of Premature Ejaculation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MorePharma Corporation (Industry)
Responsible Party: Luz Maria Lopez - Martinez MD, MorePharma Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MPEP-01
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2009-12

CONDITIONS: Premature Ejaculation
Keywords: premature ejaculation; paroxetine; daily treatment
MeSH Terms: conditions — Premature Ejaculation | interventions — Paroxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- paroxetine 15mg (Experimental): Active treatment with daily dose of paroxetine 15mg.
  Interventions: Drug: paroxetine
- paroxetine 20 mg (Experimental): Active treatment daily dose of paroxetine 20 mg
  Interventions: Drug: paroxetine
- placebo (Experimental): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: paroxetine — daily dose of paroxetine 15mg for 12 weeks
  Arms: paroxetine 15mg
Drug: paroxetine — active daily treatment with paroxetine 20 mg
  Arms: paroxetine 20 mg
Drug: placebo — active daily treatment with placebo
  Arms: placebo

SUMMARY:
As study to investigate the efficacy and safety of daily doses of paroxetine of 15 and 20 mg for the treatment of premature ejaculation

DETAILED DESCRIPTION:
Randomized, double blind, placebo controlled, prospective and parallel trial. Men with premature ejaculation using the Diagnostic and Statistical Manual of Mental Disorders, fourth edition, text revision criteria for at least 6 months, with an intravaginal ejaculatory latency time (IELT) ≤ 3 minutes. Three treatments are to be compared: placebo, 15 mg or 20 mg paroxetine for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* men between 20 and 70 years of age
* with a stable relationship with a female partner
* with the intention to continue with the same partner for the duration of the study
* with diagnosis of premature ejaculation according to the criteria established in the Diagnostic and Statistical Manual of Mental Disorders IV edition, Revised Text for at least 6 months before inclusion
* with an Intravaginal Ejaculatory Latency Time (IELT) ≤ 3 minutes in at least 75 % of a minimum of three sexual encounters, elapsing between them at least 18 hours during the selection phase of the study
* with agreement to avoid pregnancy or planned surgery during the study,
* female participants should not be pregnant at the inclusion
* both male and female partners had to agree to participate and to sign the informed consent form

Exclusion Criteria:

* any medical or surgical condition that could be associated with the initiation of premature ejaculation for secondary PE
* history of myocardial infarction or stroke in the last 6 months
* hemorrhagic disorder, hepatitis B or C, HIV infection, penile implant surgery at any time
* alcohol or drug abuse in the last 2 years
* any medical or psychiatric condition that could interfere with study procedures and evaluations
* uncontrolled diabetes
* hypotension (defined as systolic/diastolic blood pressure < 90/50 mm Hg)
* uncontrolled hypertension
* diagnosis of erectile dysfunction or a score ≤ 21 in the erectile function domain of the International Index of Erectile Function (IIEF) at inclusion
* treatment with any investigational drug in the last month or 5 times the half life of the drug
* use of medications that could enhance the effect of paroxetine,
* known intolerance to selective serotonin recapture inhibitors
* hypoactive sexual desire not caused by PE
* sexual dysfunction in the female partner that could interfere with participation
* any other significant clinical conditions that could interfere with study procedures
* employees of research sites and relatives of researchers

Ages: 20 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2008-08; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Intravaginal Ejaculatory Latency Time (IELT) | Visit 2 Baseline, Visit 3 and Visit end of treatment, at 2, 6 and 12 weeks after entry to study respectively

SECONDARY OUTCOMES:
Score of the control domain of the Index of Premature Ejaculation | Visit 1, Screening, Visit 2 Baseline, Visit 3 and Visit 4 end of treatment, at entry , 2, 6 and 12 weeks after entry to study, respectively
Score of the sexual satisfaction domain of the Index of Premature Ejaculation | Visit 1 Screening, Visit 2 Baseline, Visit 3 and Visit 4 end of treatment, Visit 1, Screening, Visit 2 Baseline, Visit 3 and Visit 4 end of treatment, at entry , 2, 6 and 12 weeks after entry to study, respectively
Score of the distress with ejaculation domain of the Index of Premature Ejaculation | Visit 1 Screning, Visit 2 Baseline, Visit 3 and Visit 4 end of treatment, Visit 1, Screening, Visit 2 Baseline, Visit 3 and Visit 4 end of treatment, at entry , 2, 6 and 12 weeks after entry to study, respectively
Erectile function domain of the International Index of Erectile Function | Visit 1 Screening, Visit 2 Baseline, Visit 3 and Viit 4 end of treatment, Visit 1, Screening, Visit 2 Baseline, Visit 3 and Visit 4 end of treatment, at entry , 2, 6 and 12 weeks after entry to study, respectively
Sexual desire domain of the International Index of Erectile Function | Visit 1 Screening,Visit 2 Baseline,Visit 3 and Visit 4 end of treatment, Visit 1, Screening, Visit 2 Baseline, Visit 3 and Visit 4 end of treatment, at entry , 2, 6 and 12 weeks after entry to study, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Eusebio Rubio-Aurioles, M.D, Ph.D., Principal Investigator — Asociacion Mexicana para la Salud Sexual, A.C.
Locations (2):
- Mexico (2):
  - Centro Especializado en Urología y Andrología del Hospital Star Médica, Mexico City, Mexico City
  - Asociacion Mexicana para la Salud Sexual, A.C., Mexico City, Mexico City

REFERENCES:
- [Background] McMahon C. Premature ejaculation: past, present, and future perspectives. J Sex Med. 2005 May;2 Suppl 2:94-5. doi: 10.1111/j.1743-6109.2005.20368.x. No abstract available. PMID 16422794
- [Background] Althof SE. Prevalence, characteristics and implications of premature ejaculation/rapid ejaculation. J Urol. 2006 Mar;175(3 Pt 1):842-8. doi: 10.1016/S0022-5347(05)00341-1. PMID 16469562
- [Background] Jannini EA, Lenzi A. Epidemiology of premature ejaculation. Curr Opin Urol. 2005 Nov;15(6):399-403. doi: 10.1097/01.mou.0000182327.79572.fd. PMID 16205491
- [Background] American Psychiatric Association: Diagnostic and Statistical Manual of Mental Disorders, 4th ed, Text Revision. Washington, DC, American Psychiatric Association, 2000.
- [Background] Waldinger MD. Towards evidence-based drug treatment research on premature ejaculation: a critical evaluation of methodology. Int J Impot Res. 2003 Oct;15(5):309-13. doi: 10.1038/sj.ijir.3901023. PMID 14562129
- [Background] Waldinger MD, Hengeveld MW, Zwinderman AH. Ejaculation-retarding properties of paroxetine in patients with primary premature ejaculation: a double-blind, randomized, dose-response study. Br J Urol. 1997 Apr;79(4):592-5. doi: 10.1046/j.1464-410x.1997.00102.x. PMID 9126089
- [Background] Waldinger MD, Zwinderman AH, Olivier B. Antidepressants and ejaculation: a double-blind, randomized, placebo-controlled, fixed-dose study with paroxetine, sertraline, and nefazodone. J Clin Psychopharmacol. 2001 Jun;21(3):293-7. doi: 10.1097/00004714-200106000-00007. PMID 11386492
- [Background] Althof S, Rosen R, Symonds T, Mundayat R, May K, Abraham L. Development and validation of a new questionnaire to assess sexual satisfaction, control, and distress associated with premature ejaculation. J Sex Med. 2006 May;3(3):465-75. doi: 10.1111/j.1743-6109.2006.00239.x. PMID 16681472
- [Background] Rosen RC, Cappelleri JC, Gendrano N 3rd. The International Index of Erectile Function (IIEF): a state-of-the-science review. Int J Impot Res. 2002 Aug;14(4):226-44. doi: 10.1038/sj.ijir.3900857. PMID 12152111